CLINICAL TRIAL: NCT04301999
Title: Clinical Effect and Safety of Photodynamic Therapy With Radiofrequency Ablation for Unresectable Extrahepatic Cholangiocarcinoma
Brief Title: Clinical Effect and Safety of PDT and RFA for Unresectable EHCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Jianfeng Yang, Deputy director of gastroenterology department, First People's Hospital of Hangzhou
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016RCB015
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Cholangiocarcinoma
Keywords: extrahepatic cholangiocarcinoma; Photodynamic therapy; radiofrequency ablation
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Photochemotherapy; 1-phenyl-3,3-dimethyltriazene; Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PDT group (Active Comparator): Patients in PDT group underwnt PDT
  Interventions: Procedure: Photodynamic therapy
- RFA group (Experimental): Patients in RFA group underwent RFA
  Interventions: Procedure: radiofrequency ablation

INTERVENTIONS:
Procedure: Photodynamic therapy — The PDT optical fiber was inserted through the dilation catheterand advanced toward the bile duct stenosis point under visualradiography. The dilation catheter was then withdrawn to leavethe PDT optical fiber directly across the stricture. Photoactivation was performed at 640 nm using a diode laser at a light dose of 180 J/cm2at power density of300 mW/cm2 and irradiation time of 600 s.
  Other Names: PDT
  Arms: PDT group
Procedure: radiofrequency ablation — an RFA electrode (Habib EndoHPB, EMcision, HitchinHerts, UK) was advanced along the guide wire into the bile duct and to the biliary stricture under X-ray fluoroscopic guidance. A 400 kHz RF generator (RITA 1500X, Angio Dynamics, USA) was connected for RFA at 7-10 W for 90 seconds.
  Other Names: RFA
  Arms: RFA group

SUMMARY:
The prognosis of patients with advanced unresectable EHCC is very poor with a median survival of 3 to 6 months. Active control of tumor growth is the key to extending stent patency and survival for patients with unresectable locally advanced EHCC. Photodynamic therapy (PDT) is by far the only modality that has shown to improve stent patency as well as over survival (OS) in patients with cholangiocarcinoma. In recent years, many studies have shown that endoscopic radiofrequency ablation (RFA) extends stent patency and possibly the survival of patients with malignant biliary obstruction. However, there are few reports comparing the clinical efficacy and advers event of these two endoscopic treatment.

DETAILED DESCRIPTION:
Extrahepatic cholangiocarcinoma (EHCC) originates from the hepatic hilar region to the lower common bile duct. The prognosis of patients with advanced unresectable EHCC is very poor with a median survival of 3 to 6 months. Active control of tumor growth is the key to extending stent patency and survival for patients with unresectable locally advanced EHCC. Photodynamic therapy (PDT) is by far the only modality that has shown to improve stent patency as well as over survival (OS) in patients with cholangiocarcinoma. In an attempt to improve stent patency placed for malignant biliary obstruction, enthusiasm for endoscopic retrograde cholangio-pancreatography (ERCP)-guided radiofrequency ablation (RFA) has been increasing in recent years. The HABIBTM EndoHBP catheter is an endoscopic bipolar RFA catheter with proven safety and effectiveness for biliary RFA of cholangiocarcinoma. Many studies have shown that endoscopic RFA extends stent patency and possibly the survival of patients with malignant biliary obstruction. However, there are few reports comparing the clinical efficacy and advers event of these two endoscopic treatment.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed cholangiocarcinoma;
* unresectable cholangiocarcinoma due to local infiltration of major vessels according to computed tomography (CT), magnetic resonance cholangiopancreatography (MRCP), or endoscopic ultrasound（EUS）;
* no previous treatment;
* adequate bone marrow and organ function (white blood cells>4.0×109/L, hemoglobin>90 g/L, and platelets>75×109/L, serum creatinine<2.0 mg/dl);
* a Karnofsky performance status (KPS) score ≥ 50;
* signed written informed consent.

Exclusion Criteria:

* imaging examination (CT, MRCP, EUS) showed distant metastasis of liver, lung and other organs;
* coexistent with other malignant tumors;
* pregnant or nursing women;
* previous gastrointestinal diversion;
* participation in another study during the month before enrollment in this study;
* alcohol and/or substance abuse or potentially poor compliance per a doctor's judgment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | two years
  OS was defined as the time from initial RFA to death or the end of the study.

SECONDARY OUTCOMES:
Adverse events | two years
  Number of patients with adverse events
Progression-free survival (PFS) | two years
  PFS was measured from randomization until the date of disease progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Yang, Principal Investigator — First People's Hospital of Hangzhou
Locations (1):
- Jianfeng Yang, Hangzhou, Zhejiang, China